CLINICAL TRIAL: NCT05163821
Title: Pilot of a New Cognitive Assessment Tool for Detecting Dementia in the Migrant Somali Population
Status: Completed | Type: Observational
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sophie Jeffery, Principal Clinical Psychologist, Greater Manchester Mental Health NHS Foundation Trust
Other Study IDs: x503s
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Somali migrants in UK, aged over 50.
  Interventions: Diagnostic Test: Manchester Somali Cognitive Assessment Tool; Diagnostic Test: ACE-III Somali Translation

INTERVENTIONS:
Diagnostic Test: Manchester Somali Cognitive Assessment Tool — Cognitive screen for dementia
Diagnostic Test: ACE-III Somali Translation — Cognitive screen for dementia

SUMMARY:
Aims

* The investigators want to find out if the tool that they have made to assess memory and thinking in Somali elders ( the 'MSCAT') is acceptable to that community and practical to administer and score.
* The public will benefit from this research because it seeks to enhance reliability of diagnosis of dementia, thus access to support and treatment for people from an ethnic minority group experiencing memory problems.

Background

* The investigators are a group of staff from the Memory Assessment Service in Manchester. There are currently no suitable tests for dementia for people from Somalia.
* Research evidence tells us there are many reasons why the tools that used now are not working. This includes: differences in culture and ways of life that are very different to a British born person who has lived in the UK for all of their life.
* Somali people find out at a later stage if they have dementia resulting in delayed treatment/support.
* This research supports the government's promise to improve the pathway to a diagnosis of dementia for minority groups.

Design and methods

* 10 participants
* The investigators will compare the assessment tool (MSCAT) that the team have developed to the Addenbrookes Cognitive Examination III tool that is typically used.
* Participants will be seen at an agreed location (e.g. home, mosque or GMMH trust site). They will meet a Somali speaking researcher to do both tests on 2 appointments and discuss how they found the tests afterwards.
* The investigators will check participants understanding of the research before they agree to take part. Verbal and written information will be provided.

Public involvement

* The local Somali community helped advise on the creation of the new MSCAT assessment tool.
* The investigators will write project information for participants in Somali and English.

Dissemination of results

• Professional conference presentations and publications

ELIGIBILITY:
Inclusion Criteria:

* The participants will all be Somali-born migrants, over the age of 50, living in the UK.

Exclusion Criteria:

* Exclusion criteria will include the presence of dementia, current delirium, or inability to complete the tasks due to visual/hearing/physical impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Somali-born migrants in UK
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Qualitative feedback on completing the cognitive screens | Immediately after completing the screen
  Interview

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester Mental Health NHS Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided